CLINICAL TRIAL: NCT00260195
Title: A School Program for Children Exposed to Violence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: RAND (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, LIsa Jaycox, Senior Behavioral Scientist, RAND
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01MH072591 (NIH); R01MH072591 (NIH); DDTR B3-PDS (Other: FDAAA)
Record Dates: First submitted 2005-11-29; First posted 2005-12-01 (Estimated); Results first posted 2014-05-22 (Estimated); Last update posted 2014-05-22 (Estimated); Status verified 2014-04

CONDITIONS: Stress Disorders, Post-Traumatic; Depression
Keywords: Trauma; Violence; Adolescent; Schools; Cognitive behavioral therapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression; Wounds and Injuries | interventions — Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- School-based cognitive behavioral support group (Experimental): Ten group lessons facilitated by a teacher or school counselor that focuses on psycho-education, development of a trauma narrative, approaching trauma-related situations, social problem solving, and cognitive skills.
  Interventions: Behavioral: School-based cognitive behavioral support group
- Wait-list control group (No Intervention): Waiting list

INTERVENTIONS:
Behavioral: School-based cognitive behavioral support group
  Other Names: Support for Students Exposed to Trauma (SSET)
  Arms: School-based cognitive behavioral support group

SUMMARY:
This study will develop a program to help school children deal with violence-related trauma.

DETAILED DESCRIPTION:
The number of children who have been indirectly or directly exposed to violence has dramatically increased in the last decade. The emotional and behavioral consequences of violence exposure can be particularly devastating to children. Interventions are needed that can reduce symptoms related to traumas already experienced and enhance children's skills for handling extreme stress that might be experienced in the future. The Cognitive-Behavioral Intervention for Trauma in Schools (CBITS) program was developed between 1998 and 2001 to help children in the Los Angeles school district deal with traumatic events. Although promising, the program required a school-based mental health clinician for implementation. This study will evaluate the effectiveness of a program adapted for the Los Angeles CBITS program that can be used by school staff in a middle school setting. The adapted CBITS program will be compared to a wait list to determine which is more effective in reducing trauma-related stress and depression among sixth grade students.

Students who have experienced violence-related trauma will be randomly assigned to receive either 10 weekly sessions of group cognitive behavioral therapy or to wait 3 months. Self-report scales and interviews will be used to assess the emotional states of participants at study entry and study completion. No follow-up visits will be required.

ELIGIBILITY:
Inclusion Criteria:

* Students in 6th and 7th grade in two participating Los Angeles area schools
* Exposure to severe violence, as either a victim or witness, within 1 year prior to study entry
* Have symptoms of post-traumatic stress disorder at study entry
* Able to speak and understand English
* Parent or guardian willing to give informed consent

Exclusion Criteria:

* Post-traumatic stress disorder symptoms that are not related to a traumatic event
* Mental retardation
* Conduct disorder that would interfere with the participant's ability to engage in group therapy

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 78 (Actual)
Dates: Start 2005-07; Primary Completion 2007-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa H. Jaycox, PhD, Principal Investigator — RAND
Locations (1):
- LAUSD Crisis Counseling and Intervention Services, LAUSD/RAND/UCLA Trauma Services Adaptation Center, Los Angeles, California, United States

REFERENCES:
- [Background] Kataoka SH, Stein BD, Jaycox LH, Wong M, Escudero P, Tu W, Zaragoza C, Fink A. A school-based mental health program for traumatized Latino immigrant children. J Am Acad Child Adolesc Psychiatry. 2003 Mar;42(3):311-8. doi: 10.1097/00004583-200303000-00011. PMID 12595784
- [Background] Stein BD, Kataoka S, Jaycox LH, Wong M, Fink A, Escudero P, Zaragoza C. Theoretical basis and program design of a school-based mental health intervention for traumatized immigrant children: a collaborative research partnership. J Behav Health Serv Res. 2002 Aug;29(3):318-26. doi: 10.1007/BF02287371. PMID 12216375
- [Background] Stein BD, Jaycox LH, Kataoka SH, Wong M, Tu W, Elliott MN, Fink A. A mental health intervention for schoolchildren exposed to violence: a randomized controlled trial. JAMA. 2003 Aug 6;290(5):603-11. doi: 10.1001/jama.290.5.603. PMID 12902363
- [Background] Jaycox LH, Stein BD, Kataoka SH, Wong M, Fink A, Escudero P, Zaragoza C. Violence exposure, posttraumatic stress disorder, and depressive symptoms among recent immigrant schoolchildren. J Am Acad Child Adolesc Psychiatry. 2002 Sep;41(9):1104-10. doi: 10.1097/00004583-200209000-00011. PMID 12218432

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We recruited and screened 6th and 7th grade students in two schools over two school years (2005-2006 and 2006-2007) in Los Angeles Unified School District.
Pre-assignment Details: There are 3 steps in enrollment: consent for screening, screening, consent for participation for those who screened positive. 383 students were screened, 193 screened positive, 78 consented for the project (active parental consent and child assent). 2 students withdrew from the school prior groups and thus did not participate further.
Groups:
- Wait-list Control Group: Students assigned to this group waited while the experimental arm received SSET, and then completed the first follow-up assessment. They then received SSET between the first and second follow-up assessment.
Period: Overall Study
Arm/Group | School-based Cognitive Behavioral Support Group | Wait-list Control Group
Started | 39 | 37
Completed | 39 | 37
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | School-based Cognitive Behavioral Support Group | Wait-list Control Group | Total
Number analyzed (Participants) | 39 | 37 | 76
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 39 | 37 | 76
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.4 (0.6) | 11.5 (0.7) | 11.5 (0.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 18 | 39
  Male | 18 | 19 | 37
Region of Enrollment [Number; unit: participants]
  United States | 39 | 37 | 76

OUTCOME MEASURES:

1. Primary Outcome: Post-traumatic Stress Disorder Symptoms
Description: We used the Child PTSD Symptom Scale (CPSS; Foa,Treadwell, Johnson, & Feeny, 2001), to assess PTSD symptoms for both screening into the program and for use in examining child outcomes over time. This scale has been used in school aged children as young as 8 and has shown good convergent and discriminant validity and high reliability (Foa et al., 2001). In our earlier work, scale internal consistency was high (Cronbach's alpha = 0.89; Jaycox et al., 2002). In this study, we use it as a continuous scale as designed, and also use cut-points to determine eligibility for the study as in prior work (Kataoka et al., 2003; Stein et al., 2003), requiring a total score of 11 or greater, indicating moderate levels of current PTSD symptoms. A high score indicates more symptoms, and total scores can range from 0 to 51.
Time Frame: Symptoms over the past two weeks were assessed at baseline, after intervention for the SSET group (10 weeks), and after all receive intervention (20 weeks).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | School-based Cognitive Behavioral Support Group | Wait-list Control Group
Number analyzed (Participants) | 39 | 37
units on a scale
  Baseline | 17.46 (10.37) | 19.41 (10.00)
  After Intervention for SSET Group | 13.72 (8.43) | 18.32 (11.31)
  After all receive intervention | 11.97 (9.07) | 15.59 (9.42)

2. Primary Outcome: Depressive Symptoms
Description: Children's Depression Inventory (CDI; Kovacs, 1981) This 27-item measure assesses children's cognitive, affective, and behavioral depressive symptoms. The scale has high internal consistency, moderate test-retest reliability, and correlates in the expected direction with measures of related constructs (e.g., self-esteem, negative attributions, and hopelessness; Kendall, Cantwell, & Kazdin, 1989). Normative data are available (Finch, Saylor, & Edwards, 1985). We used a 26-item version of the scale that omits an item about suicidal ideation. Higher scores indicate more symptoms, and total scores can range from 0 to 52.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | School-based Cognitive Behavioral Support Group | Wait-list Control Group
Number analyzed (Participants) | 39 | 37
units on a scale
  Baseline | 13.87 (8.52) | 14.32 (9.20)
  After Intervention for SSET Group | 11.77 (7.90) | 14.92 (9.02)
  After all receive intervention | 12.21 (9.79) | 12.91 (8.55)

3. Primary Outcome: Parent Report of Behavioral Problems
Description: Strengths and Difficulties Questionnaire-Parent Report, and Teacher Report (SDQ, Goodman, 1997; Goodman, Meltzer, & Bailey, 1998) This questionnaire contains 25 items, 20 assessing problem areas (emotional symptoms, conduct problems, hyperactivity/inattention, and peer relationship problems), 5 assessing prosocial behavior, and items that tap functional impairment related to these problems (Goodman, 1999). Higher scores indicate more problems, with total scores for problem areas ranging from 0 to 40.
Time Frame: Problems over the prior month were assessed at baseline, after intervention for the SSET group (10 weeks), and after all receive intervention (20 weeks).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | School-based Cognitive Behavioral Support Group | Wait-list Control Group
Number analyzed (Participants) | 39 | 37
units on a scale
  Baseline | 11.64 (5.80) | 12.46 (5.90)
  After Intervention for SSET Group | 9.72 (4.94) | 11.30 (5.84)
  After all receive intervention | 8.41 (4.91) | 8.91 (6.08)

4. Primary Outcome: Teacher Report of Behavior Problems
Description: Strengths and Difficulties Questionnaire-Parent Report, and Teacher Report (SDQ, Goodman, 1997; Goodman, Meltzer, & Bailey, 1998) This questionnaire contains 25 items, 20 assessing problem areas (emotional symptoms, conduct problems, hyperactivity/inattention, and peer relationship problems), 5 assessing prosocial behavior, and items that tap functional impairment related to these problems (Goodman, 1999). Higher scores indicates more problems, with total problem area scores ranging from 0 to 40.
Time Frame: Problems over the month were assessed at baseline, after intervention for the SSET group (10 weeks), and after all receive intervention (20 weeks).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | School-based Cognitive Behavioral Support Group | Wait-list Control Group
Number analyzed (Participants) | 39 | 37
units on a scale
  Baseline | 11.33 (7.87) | 8.59 (7.37)
  After Intervention for SSET Group | 10.28 (6.95) | 9.30 (7.98)
  After all receive intervention | 10.47 (5.75) | 9.19 (6.86)

ADVERSE EVENTS:
Time Frame: One school year (from screening through last follow-up)
Arm/Group | School-based Cognitive Behavioral Support Group | Wait-list Control Group
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/37
Other Adverse Events (participants affected / at risk) | 0/39 | 0/37

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No